CLINICAL TRIAL: NCT00668161
Title: Exercise Intervention Trial for Colorectal Polyp Patients
Brief Title: Effect of Exercise on Biomarkers of Colon Cancer Risk
Acronym: APPEAL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Anne McTiernan, MD, PhD, Fred Hutchinson Cancer Research Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: APPEAL CA77572-01; FHCRC-4838, R01 CA77572-01
Record Dates: First submitted 2008-04-24; First posted 2008-04-29 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Colon Cancer Prevention
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Exercise
  Interventions: Behavioral: Exercise
- 2 (No Intervention): Control

INTERVENTIONS:
Behavioral: Exercise — 60 minutes/session of aerobic exercise, 6 d/week at 50-50% HHR. All sessions will begin with 10 minutes of stretching and 5 minutes of warm-up, and will end with 5 minutes of cool down.
  Arms: 1

SUMMARY:
There is strong observational epidemiologic evidence that physical activity is inversely associated with risk of colon cancer occurrence in both men and women. This association has been found in over 30 observational studies, and appears to be independent of effects of diet, body fat mass, and other potential confounding factors. Prior to large-scale recommendations regarding exercise as a means of preventing colon cancer, however, more information is needed regarding the type of exercise, when it must be initiated, and how much must be done, in order to produce a protective effect. Information on the mechanisms and biological pathways through which exercise might protect the colon will aid in developing the answers to these questions.

This is a randomized controlled trial of a one-year moderate/vigorous exercise intervention vs. delayed- exercise control on various biomarkers of colon cancer risk in persons that have undergone a colonoscopy within the past 36 months.. The trial is designed to establish the effects of the exercise intervention on colorectal cell proliferation and terminal differentiation, and on factors that may lie in the pathway between exercise and proliferation and apoptosis, in colon and rectal epithelium. It will provide data on: 1) the efficacy of a one-year moderate intensity aerobic exercise program in modulating these processes to a pattern considered low risk for colon cancer, and 2) the mechanisms whereby exercise may lower colon cancer risk in humans. To the investigators' knowledge, this will be the first study of its kind.

DETAILED DESCRIPTION:
The specific aims of the proposed study are:

1. To measure the effects of a one-year moderate/vigorous intensity aerobic exercise program vs. a delayed-exercise control program in persons that have undergone a colonoscopy within the past 36 months on proliferation rate in the upper part of colon and rectal mucosa crypts.
2. To also measure the effects of a one-year moderate/vigorous intensity aerobic exercise program vs. delayed-exercise control program in persons that have undergone a colonoscopy within the past 36 months on:

   * expression of apoptosis-related proteins (bax/bcl-2 ratio) in colon and rectal mucosal biopsies
   * rectal mucosal prostaglandin levels
   * fasting serum/plasma insulin, glucose, triglycerides, insulin-like growth factor 1(IGF-1), and IGF binding protein-3 (IGFPB-3)
   * body fat mass and distribution (body mass index, waist and hip circumferences, bioelectrical impedance, DEXA scan)
   * subcutaneous abdominal and intra-abdominal fat mass (measured by one-slice CT scan at the L4 level)
   * fitness (VO2max)
   * quality of life (measured by standardized self-report instruments)
   * sleep quality

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Completed a colonoscopy within the past 36 months
* Ages 40-75 years at time of identification
* Sedentary activity pattern
* Gives informed consent, agrees to be randomly assigned
* Able to perform all study requirements, able to follow directions and complete forms

Exclusion Criteria:

* Colorectal cancer at any time; any other invasive cancer within the past 10 years (simple basal or squamous cell carcinoma okay)
* Plans to leave Western Washington during the follow-up period
* Morbidly obese (BMI > 41), weight loss of > 10 pounds in the previous 3 months
* Familial polyposis, Gardner's syndrome, or other known familial colorectal cancer syndrome
* Ulcerative colitis or short bowel
* "Excessive"(> 3 x week) laxative or enema use that might interfere with rectal crypt studies
* Current use of certain medications likely to interfere with success of the intervention, or with outcomes measures (for example, anticoagulants because of risk from colorectal biopsy, diet medications within past 6 months)
* Diabetes mellitus or fasting glucose > 140
* Hemochromatosis- if diagnosed by physician
* Abnormal screening labs (hematocrit < 32 or > 48, white blood cells < 3.0 or > 15.0, potassium < 3.5 or > 5.3, fasting glucose > 140, creatinine > 2.0), or abnormalities on screening physical exam judged by study physicians to contraindicate participation in an exercise program
* Contraindications for entry into a training program 131 including: unstable angina, uncontrolled hypertension (systolic > 200, diastolic > 100), orthostatic hypotension (>20 mm fall in systolic), moderate/severe aortic stenosis, uncontrolled arrhythmia, uncontrolled congestive heart failure, third degree heart block, pericarditis, myocarditis, pulmonary/systemic embolism within the past 6 months, thrombophlebitis, ST displacement > 3 mm at rest, history of cardiac arrest)
* Contraindications for exercise testing 131 including: recent (within 6 months) cardiac event (MI, pulmonary edema, myocarditis, pericarditis), unstable angina, uncontrolled arrhythmia, third degree heart block, left bundle branch block, acute congestive failure, recent (within 6 months) pulmonary/systemic embolus, severe electrolyte abnormality
* Meets criteria to stop screening exercise test 131 as decided by overseeing physician
* Volunteering in order to lose weight; alcohol or drug abuse, significant mental or emotional problems such as would interfere with compliance (as assessed by study staff impression)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2001-01; Primary Completion 2004-12 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Proliferation rate in the upper part of colon and rectal mucosa crypts. | Baseline and 12-months

SECONDARY OUTCOMES:
expression of apoptosis-related proteins (bax/bcl-2 ratio) in colon and rectal mucosal biopsies | Baseline and 12-months
rectal mucosal prostaglandin levels | baseline and 12-months
fasting serum/plasma insulin, glucose, triglycerides, insulin-like growth factor 1(IGF-1), and IGF binding protein-3 (IGFPB-3) | baseline and 12-months
body fat mass and distribution (body mass index, waist and hip circumferences, bioelectrical impedance, DEXA scan)and subcutaneous abdominal and intra-abdominal fat mass (measured by one-slice CT scan at the L4 level) | baseline and 12-months
quality of life (measured by standardized self-report instruments) and sleep quality | baseline and 12-months

CONTACTS AND LOCATIONS:
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Result] Hawkins VN, Foster-Schubert K, Chubak J, Sorensen B, Ulrich CM, Stancyzk FZ, Plymate S, Stanford J, White E, Potter JD, McTiernan A. Effect of exercise on serum sex hormones in men: a 12-month randomized clinical trial. Med Sci Sports Exerc. 2008 Feb;40(2):223-33. doi: 10.1249/mss.0b013e31815bbba9. PMID 18202581
- [Result] Abrahamson PE, King IB, Ulrich CM, Rudolph RE, Irwin ML, Yasui Y, Surawicz C, Lampe JW, Lampe PD, Morgan A, Sorensen BE, Ayub K, Potter JD, McTiernan A. No effect of exercise on colon mucosal prostaglandin concentrations: a 12-month randomized controlled trial. Cancer Epidemiol Biomarkers Prev. 2007 Nov;16(11):2351-6. doi: 10.1158/1055-9965.EPI-07-0120. PMID 18006923
- [Result] Campbell KL, McTiernan A, Li SS, Sorensen BE, Yasui Y, Lampe JW, King IB, Ulrich CM, Rudolph RE, Irwin ML, Surawicz C, Ayub K, Potter JD, Lampe PD. Effect of a 12-month exercise intervention on the apoptotic regulating proteins Bax and Bcl-2 in colon crypts: a randomized controlled trial. Cancer Epidemiol Biomarkers Prev. 2007 Sep;16(9):1767-74. doi: 10.1158/1055-9965.EPI-07-0291. PMID 17855695
- [Result] McTiernan A, Sorensen B, Irwin ML, Morgan A, Yasui Y, Rudolph RE, Surawicz C, Lampe JW, Lampe PD, Ayub K, Potter JD. Exercise effect on weight and body fat in men and women. Obesity (Silver Spring). 2007 Jun;15(6):1496-512. doi: 10.1038/oby.2007.178. PMID 17557987
- [Result] McTiernan A, Yasui Y, Sorensen B, Irwin ML, Morgan A, Rudolph RE, Surawicz C, Lampe JW, Ayub K, Potter JD, Lampe PD. Effect of a 12-month exercise intervention on patterns of cellular proliferation in colonic crypts: a randomized controlled trial. Cancer Epidemiol Biomarkers Prev. 2006 Sep;15(9):1588-97. doi: 10.1158/1055-9965.EPI-06-0223. PMID 16985018
- [Derived] Duggan C, Yu M, Willbanks AR, Tapsoba JD, Wang CY, Grady WM, McTiernan A. Exercise effects on DNA methylation in EVL, CDKN2A (p14, ARF), and ESR1 in colon tissue from healthy men and women. Epigenetics. 2022 Oct;17(10):1070-1079. doi: 10.1080/15592294.2021.1982512. Epub 2021 Oct 6. PMID 34550860
- [Derived] Imayama I, Alfano CM, Mason CE, Wang C, Xiao L, Duggan C, Campbell KL, Foster-Schubert KE, Wang CY, McTiernan A. Exercise adherence, cardiopulmonary fitness and anthropometric changes improve exercise self-efficacy and health-related quality of life. J Phys Act Health. 2013 Jul;10(5):676-89. doi: 10.1123/jpah.10.5.676. Epub 2012 Oct 4. PMID 23036856
- [Derived] Campbell K, Foster-Schubert K, Xiao L, Alfano C, Bertram LC, Duggan C, Irwin M, McTiernan A. Injuries in sedentary individuals enrolled in a 12-month, randomized, controlled, exercise trial. J Phys Act Health. 2012 Feb;9(2):198-207. doi: 10.1123/jpah.9.2.198. PMID 22368219
- [Derived] Imayama I, Alfano CM, Cadmus Bertram LA, Wang C, Xiao L, Duggan C, Campbell KL, Foster-Schubert KE, McTiernan A. Effects of 12-month exercise on health-related quality of life: a randomized controlled trial. Prev Med. 2011 May;52(5):344-51. doi: 10.1016/j.ypmed.2011.02.016. Epub 2011 Mar 1. PMID 21371498